CLINICAL TRIAL: NCT02719782
Title: A Phase I Study T Cell Receptor-Redirected T Cells Infusions in Subjects With Recurrent HBV-Related Hepatocellular Carcinoma in Post Liver Transplantation
Brief Title: A Study of TCR-Redirected T Cell Infusion in Subject With Recurrent HBV-related HCC Post Liver Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lion TCR Pte. Ltd. (Industry)
Collaborators: Agency for Science, Technology and Research (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-2-1
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Recurrent Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBV/TCR T cell Infusion (Experimental): This is a single-arm study.
  Patients will receive a total of 2 cycles, in which first 28-day treatment cycle consists of escalating doses of TCR-T on Day 1, Day 8, Day 15 and Day 22, followed by every 2-week dosing on Day 1, Day 15, Day 29 and Day 43 of second (final) cycle. A one month treatment break will be given between the cycles.
  Interventions: Biological: Biological: TCR-T

INTERVENTIONS:
Biological: Biological: TCR-T — Autologous T cells transfected with mRNA encoding HBV antigen-specific TCR

SUMMARY:
Hepatocellular carcinoma (HCC) recurrence rate is high among liver transplant patients, while treatment measures are limited. This study plans to recruit 10 patients with Hepatitis B virus (HBV) related HCC who underwent liver transplantation and are confirmed to have recurrent HCC. The objective of the study is to assess the safety, tolerability and effectiveness of the HBV specific T cell receptor (HBV/TCR) redirected T cell in the target population.

DETAILED DESCRIPTION:
This is a phase I, single armed and open labelled trial in patients with recurrent HBV related HCC after liver transplantation. Subjects who meet eligibility criteria will receive escalating doses of HBV specific T cell receptor (TCR-T) on Day 1, Day 8, Day 15 and Day 22 of the first 28-day treatment cycle, followed by every 2-week dosing on Day 1, Day 15, Day 29 and Day 43 of repeated cycle. A 21-day treatment break will be given between each cycle. Treatment will be continued until disease progression unless otherwise specified per investigator's discretion. Subjects will be followed up post treatment for safety monitoring, including monthly follow up for the first three month and every 2-monthly follow up up to 24 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as hepatocellular carcinoma (HCC)
* Underwent liver transplantation and confirmed recurrent HCC post operation
* Seropositive for hepatitis B surface antigen
* No major post-operative complication
* Life expectancy of at least 12 weeks
* Ability to provide informed consent
* Ability to comply with study procedures
* HLA profile matching with HLA-class I restriction element of the available T cell receptors

Exclusion Criteria:

* Administration of any other cell therapy, including NK, CIK, DC, CTL, CAR-T, stem cells or combined therapy of the kind within 3 months prior to enrolment
* Second primary malignancy that is clinically detectable at the time of consideration for study enrolment
* Likelihood to require steroid treatment during the period of the clinical trial
* Any other concurrent liver infections such as hepatitis A, C or D infection
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumours including metastatic brain disease.
* Any condition that is unstable or which could jeopardise the safety of the patient and his/her compliance in the study
* Patients with reproductive potential who tested positive for serum or urine pregnancy test result within 14 days prior to enrolment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07-02 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the TCR-T treatment | Start of treament until 1 month after last treatment

SECONDARY OUTCOMES:
Efficacy of induction of tumor specific T cell responses as measured by the persistence of HBV specific T cells in peripheral blood samples at several time points following adoptive transfer | Start of treatment until disease progression, and subsequent follow up up to 24 months post treatment
Systemic release of inflammatory cytokines after administration of transduced T cells compared to baseline | Start of treatment until disease progression, and subsequent follow up up to 24 months post treatment

OTHER OUTCOMES:
1-year PFS (progression free survival) which is measured by the number of patients with stable disease after 1 year, using mRECIST | Start of treatment until disease progression, median 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhang, MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University; Antonio Bertoletti, MD, Study Chair — Duke-NUS Graduate Medical School
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qasim W, Brunetto M, Gehring AJ, Xue SA, Schurich A, Khakpoor A, Zhan H, Ciccorossi P, Gilmour K, Cavallone D, Moriconi F, Farzhenah F, Mazzoni A, Chan L, Morris E, Thrasher A, Maini MK, Bonino F, Stauss H, Bertoletti A. Immunotherapy of HCC metastases with autologous T cell receptor redirected T cells, targeting HBsAg in a liver transplant patient. J Hepatol. 2015 Feb;62(2):486-91. doi: 10.1016/j.jhep.2014.10.001. Epub 2014 Oct 13. PMID 25308176
- [Background] Gehring AJ, Xue SA, Ho ZZ, Teoh D, Ruedl C, Chia A, Koh S, Lim SG, Maini MK, Stauss H, Bertoletti A. Engineering virus-specific T cells that target HBV infected hepatocytes and hepatocellular carcinoma cell lines. J Hepatol. 2011 Jul;55(1):103-10. doi: 10.1016/j.jhep.2010.10.025. Epub 2010 Nov 23. PMID 21145860
- [Background] Koh S, Shimasaki N, Suwanarusk R, Ho ZZ, Chia A, Banu N, Howland SW, Ong AS, Gehring AJ, Stauss H, Renia L, Sallberg M, Campana D, Bertoletti A. A practical approach to immunotherapy of hepatocellular carcinoma using T cells redirected against hepatitis B virus. Mol Ther Nucleic Acids. 2013 Aug 13;2(8):e114. doi: 10.1038/mtna.2013.43. PMID 23941866
- [Derived] Yang F, Zheng X, Koh S, Lu J, Cheng J, Li P, Du C, Chen Y, Chen X, Yang L, Chen W, Wong RW, Wai LE, Wang T, Zhang Q, Chen W. Messenger RNA electroporated hepatitis B virus (HBV) antigen-specific T cell receptor (TCR) redirected T cell therapy is well-tolerated in patients with recurrent HBV-related hepatocellular carcinoma post-liver transplantation: results from a phase I trial. Hepatol Int. 2023 Aug;17(4):850-859. doi: 10.1007/s12072-023-10524-x. Epub 2023 Apr 17. PMID 37067675